CLINICAL TRIAL: NCT01470326
Title: Viviant®20mg Special Investigation (Regulatory Post Marketing Commitment Plan)
Brief Title: Viviant 20mg Special Investigation (Regulatory Post Marketing Commitment Plan)
Acronym: VIOLINE
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1781007
Record Dates: First submitted 2011-11-09; First posted 2011-11-11 (Estimated); Results first posted 2018-11-05 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-03

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Post menopausal women; SERM; Japanese; Viviant; Regulatory Post Marketing Commitment Plan; Long term treatment
MeSH Terms: conditions — Osteoporosis | interventions — bazedoxifene

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bazedoxifene Tablets: Subjects taking Bazedoxifene Tablets
  Interventions: Drug: Bazedoxifene

INTERVENTIONS:
Drug: Bazedoxifene — For adults, take 1 tablet (20 mg of the active ingredient) at a time, once a day.

SUMMARY:
In this survey, to collect the safety and efficacy information of Bazedoxifene in daily medical practice will be examined. In addition, the necessity of special Investigation and post-marketing clinical studies will be examined, while investigating unexpected adverse drug reactions during the survey period and understanding of the status of frequency of adverse drug reactions in daily medical practice.

DETAILED DESCRIPTION:
All the subjects whom an investigator prescribes the first Bazedoxifene (Viviant) Tablets should be registered consecutively until the number of subjects reaches target number in order to extract patients enrolled into the investigation at random.

ELIGIBILITY:
Inclusion Criteria:

* Post menopausal women subjects with Osteoporosis who has no experience of use of Bazedoxifene.

Exclusion Criteria:

* Subject with present or past venous thromboembolism such as deep venous thrombosis, pulmonary embolism, or retinal venous thrombosis
* Subject in long-term immovability (postoperative recovery, long-term bed rest)
* Subject with antiphospholipid antibody syndrome

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: The subjects whom an investigator involving B1781007 prescribes the Bazedoxifene Tablets.
Sampling Method: Probability Sample
Enrollment: 3187 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1781007&StudyName=Viviant%2020mg%20Special%20Investigation%20%28Regulatory%20Post%20Marketing%20Commitment%20Plan%29%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Viviant (Bazedoxifene Acetate): Participants who received Viviant as indicated in the approved local product document were observed for a period of 3 years. The dosage can be adjusted as per physician's discretion.
Period: Overall Study
Arm/Group | Viviant (Bazedoxifene Acetate)
Started | 3187
Completed | 3034
Not Completed | 153
Not completed — Protocol Violation | 32
Not completed — No Drug Administration Information | 2
Not completed — No Visit After 1st Day of Treatment | 119

BASELINE CHARACTERISTICS:
Arm/Group | Viviant (Bazedoxifene Acetate)
Number analyzed (Participants) | 3034
Age, Customized [Count of Participants; unit: Participants]
  <15 years | 0
  ≥15 and <65 years | 514
  ≥65 years | 2520
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3034
  Male | 0
Smoking Status [Count of Participants; unit: Participants]
  Smoker | 94
  Non-Smoker | 2211
  Unknown | 729
Use of Steroid [Count of Participants; unit: Participants]
  Yes | 101
  No | 2523
  Unknown | 410
Use of Previous Medication [Count of Participants; unit: Participants]
  Yes | 1271
  No | 1647
  Unknown | 116
Use of Concomitant Medication [Count of Participants; unit: Participants]
  Yes | 2103
  No | 931
Fracture History [Count of Participants; unit: Participants]
  Yes | 842
  No | 1807
  Unknown | 385

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Related Adverse Events
Description: A treatment-related adverse event was any untoward medical occurrence attributed to Viviant in a participant who received Viviant. A treatment-related serious adverse event was a treatment-related adverse event resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; lifethreatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Relatedness to Viviant was assessed by the physician.
Time Frame: 3 years
Population: The safety analysis set comprised of participants who satisfied the inclusion criteria and had received Viviant at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | Viviant (Bazedoxifene Acetate)
Number analyzed (Participants) | 3034
Participants
  Treatment-related Adverse Event | 137
  Treatment-related Serious Adverse Event | 5

2. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events Unexpected From Japanese Package Insert
Description: A treatment-related adverse event was any untoward medical occurrence attributed to Viviant in a participant who received Viviant. Expectedness of the adverse event was determined according to the Japanese package insert. Relatedness to Viviant was assessed by the physician.
Time Frame: 3 years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Viviant (Bazedoxifene Acetate)
Number analyzed (Participants) | 3034
Participants | 80

3. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events by Age
Description: A treatment-related adverse event was any untoward medical occurrence attributed to Viviant in a participant who received Viviant. Relatedness to Viviant was assessed by the physician. Participants with treatment-related adverse events were counted by age to assess whether it was a risk factor for the occurrence of treatment-related adverse events.
Time Frame: 3 years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Viviant (Bazedoxifene Acetate)
Number analyzed (Participants) | 3034
Participants
  <15 years: number analyzed (Participants) | 0
  ≥15 and <65 years: number analyzed (Participants) | 514
  ≥15 and <65 years | 25
  ≥65 years: number analyzed (Participants) | 2520
  ≥65 years | 112

4. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events by Smoking Status
Description: A treatment-related adverse event was any untoward medical occurrence attributed to Viviant in a participant who received Viviant. Relatedness to Viviant was assessed by the physician. Participants with treatment related-adverse events were counted by smoking status to assess whether it was a risk factor for the occurrence of treatment-related adverse events.
Time Frame: 3 years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Viviant (Bazedoxifene Acetate)
Number analyzed (Participants) | 3034
Participants
  Smoker: number analyzed (Participants) | 94
  Smoker | 0
  Non-Smonker: number analyzed (Participants) | 2211
  Non-Smonker | 85
  Unknown: number analyzed (Participants) | 729
  Unknown | 52

5. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events by Use of Steroid
Description: A treatment-related adverse event was any untoward medical occurrence attributed to Viviant in a participant who received Viviant. Relatedness to Viviant was assessed by the physician. Participants with treatment-related adverse events were counted by the use of steroid to assess whether it was a risk factor for the occurrence of treatment-related adverse events.
Time Frame: 3 years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Viviant (Bazedoxifene Acetate)
Number analyzed (Participants) | 3034
Participants
  Yes: number analyzed (Participants) | 101
  Yes | 13
  No: number analyzed (Participants) | 2523
  No | 99
  Unknown: number analyzed (Participants) | 410
  Unknown | 25

6. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events by Use of Previous Medication
Description: A treatment-related adverse event was any untoward medical occurrence attributed to Viviant in a participant who received Viviant. Relatedness to Viviant was assessed by the physician. Participants with treatment-related adverse events were counted by the use of previous medications to assess whether they were risk factors for the occurrence of treatment-related adverse events.
Time Frame: 3 years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Viviant (Bazedoxifene Acetate)
Number analyzed (Participants) | 3034
Participants
  Yes: number analyzed (Participants) | 1271
  Yes | 66
  No: number analyzed (Participants) | 1647
  No | 64
  Unknown: number analyzed (Participants) | 116
  Unknown | 7

7. Primary Outcome: Number of Participants With Any Fracture
Description: Occurrence of any fracture after Viviant administration was examined to evaluate effectiveness of Viviant. The event of fracture was defined as an event which included "fracture" in Preferred Term (PT) or Lowest Level Term (LLT) of the MedDRA/J version 18.1.
Time Frame: 3 years
Population: The effectiveness analysis set was identical with the safety analysis set which comprised of participants who satisfied the inclusion criteria and had received Viviant at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | Viviant (Bazedoxifene Acetate)
Number analyzed (Participants) | 3034
Participants | 53

8. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events by Use of Concomitant Medication
Description: A treatment-related adverse event was any untoward medical occurrence attributed to Viviant in a participant who received Viviant. Relatedness to Viviant was assessed by the physician. Participants with treatment-related adverse events were counted by the use concomitant medications to assess whether they were risk factors for the occurrence of treatment-related adverse events.
Time Frame: 3 years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Viviant (Bazedoxifene Acetate)
Number analyzed (Participants) | 3034
Participants
  Yes: number analyzed (Participants) | 2098
  Yes | 101
  No: number analyzed (Participants) | 936
  No | 36

ADVERSE EVENTS:
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both serious and nonserious events during the study.
Arm/Group | Viviant (Bazedoxifene Acetate)
Serious Adverse Events (participants affected / at risk) | 95/3034
Other Adverse Events (participants affected / at risk) | 83/3034
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Viviant (Bazedoxifene Acetate) (N=3034)
Biliary tract infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm recurrence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anaemia (Blood and lymphatic system disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Marasmus (Metabolism and nutrition disorders) | 1
Altered state of consciousness (Nervous system disorders) | 1
Cerebellar infarction (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 5
Hepatic encephalopathy (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Atrioventricular block complete (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 4
Cardiac failure acute (Cardiac disorders) | 4
Cardiac failure congestive (Cardiac disorders) | 1
Cardiac failure chronic (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Aortic dissection (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 4
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2
Anorectal disorder (Gastrointestinal disorders) | 1
Autoimmune pancreatitis (Gastrointestinal disorders) | 1
Colitis ischaemic (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Bile duct obstruction (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Calculus ureteric (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Condition aggravated (General disorders) | 2
Death (General disorders) | 4
Disease progression (General disorders) | 1
Haemoglobin decreased (Investigations) | 1
Bone contusion (Injury, poisoning and procedural complications) | 1
Compression fracture (Injury, poisoning and procedural complications) | 3
Fall (Injury, poisoning and procedural complications) | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 5
Femur fracture (Injury, poisoning and procedural complications) | 5
Fracture (Injury, poisoning and procedural complications) | 2
Heat illness (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 5
Radius fracture (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Viviant (Bazedoxifene Acetate) (N=3034)
Back pain (Musculoskeletal and connective tissue disorders) | 25
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 18
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 20
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.